CLINICAL TRIAL: NCT06865547
Title: ProA Study: ProActive Management Model in Metastatic Hormone Sensitive Prostate Cancer (mHSPC) Treated by Apalutamide
Acronym: ProA
Status: Enrolling by invitation | Type: Observational
Sponsor: Yonghong Li (Other)
Responsible Party: Sponsor-Investigator, Yonghong Li, Chief physician, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2024-FXY-317
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer (Adenocarcinoma)
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: The 4A ProActive Management Model — This model focuses on four key areas - Active Education, Active Prevention Strategies, Active Management, and Active Follow-up. Active Education involves providing patients with detailed information on treatment regimens, potential AEs, and self-care through verbal education, reminder cards, and direct counseling. Active Prevention Strategies aims to directly reduce risks through nursing care bundles that incorporate supportive medications, fall risk assessments, and dietary guidance. Active Management establishes robust protocols for early AE reporting, rapid treatment, and standardized order sets. Active Follow-up comprises additional outpatient visits, patient surveys, medication refill coordination, and pharmacist/nurse follow-up calls to closely monitor patient adherence and symptoms.

SUMMARY:
This is a Phase 4, multi-center, single arm, open-label clinical study to evaluate whether participants with mHSPC treated with apalutamide will benefit from the 4A ProActive Management Model.

The study will include a Screening Period of up to 14 days before assignment on Day 1 to establish study eligibility. Participants will get 4A ProActive Management according to the protocol .

As the background disease treatment, participants will received apalutamide according to local label (240 mg, 4 × 60 mg tablets, orally once daily with or without food) with duration of at least 6 months. Participants will have a Safety Follow-Up Visit within 30 days after the Visit 7.

Participants will be monitored for safety, starting from the time of signing the informed consent until 30 days after the Visit 7. AEs including laboratory AEs will be graded and summarized using Version 5.0 of the National Cancer Institute Common Terminology Criteria for Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be a man ≥ 18 years of age, at the time of signing the informed consent.
2. Participants who are diagnosed of prostate adenocarcinoma as confirmed by the Investigator and intend to be prescribed by apalutamide.
3. Androgen deprivation therapy (ie, medical or surgical castration) must have been started less than 3 months prior to screening.
4. Participant will be initiated with apalutamide and androgen deprivation therapy.
5. Have an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1. Participants with ECOG PS 2 or 3 are eligible for the study if the ECOG PS score is related to stable physical limitations (eg, wheelchair-bound due to prior spinal cord injury) and not related to prostate cancer or associated therapy.
6. Be able to swallow whole apalutamide tablets.
7. A participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person during the study and for at least 3 months after receiving the last dose of apalutamide.

   If the participant's partner is a person of childbearing potential, the participant must use condoms (with or without spermicide) and the sexual partner of the participant must also be practicing a highly effective method of contraception where conception is possible. A vasectomized participant must still use a condom (with or without spermicide) and the partner is also required to use a highly effective method of contraception where conception is possible.
8. A participant must agree not to donate sperm for the purposes of reproduction during the study and for at least 3 months after receiving the last dose of apalutamide. If applicable, participants should consider preservation of sperm prior to study treatment as anti cancer treatments may impair fertility.
9. A participant must agree not to plan to conceive a child while enrolled in this study or within 3 months after the last dose of apalutamide.
10. Participants are capable of giving signed informed consent.

Exclusion Criteria:

1. Pathological findings consistent with small cell, ductal or neuroendocrine carcinoma of the prostate.
2. Participant has active (new or progressive) brain metastases for whom the treating physician determines that central nervous system (CNS) specific treatment is required immediately or during the first cycle of therapy. Lymph nodes as only sites of metastases.

   Those with active (new or progressive) brain metastases for whom the treating physician determines that CNS specific treatment is not required immediately or during the first cycle of therapy are eligible for inclusion.
3. Visceral (ie, liver or lung) metastases as only sites of metastases.
4. Current evidence of any of the following:

   1. Any of the following within 6 months prior to first dose of apalutamide: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, uncontrolled hypertension, clinically significant arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias or New York Heart Association Class II to IV heart disease.
   2. Gastrointestinal disorder affecting absorption.
   3. Active infection requiring systemic therapy such as human immunodeficiency virus.
   4. Active or symptomatic viral hepatitis or chronic liver disease; ascites or bleeding disorders secondary to hepatic dysfunction
5. History of seizure or known condition that has been determined to significantly predispose to seizure per Investigator (including, but not limited to, loss of consciousness within 1 year prior to screening, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect).
6. Participant have known allergies, hypersensitivity, or intolerance to apalutamide or its excipients (please refer to Investigator's Brochure).
7. Prior novel hormone therapy or chemotherapy.
8. Treatment with drugs known to lower the seizure threshold within 4 weeks prior to enrollment.
9. Current or prior treatment with anti-epileptic medications for the treatment of seizures.
10. Administration of other investigational therapeutic agents, blood product support, growth factor support or invasive surgical procedure (not including surgical castration) ≤ 28 days prior to the first dose of apalutamide or currently enrolled in an investigational study.
11. Any condition or situation that in the opinion of the Investigator, would preclude participation in the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants with mHSPC treated with apalutamide
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the change of FACT-P total score after 6 months from baseline.The Fact-P is the Functional Assessment of Cancer Therapy-Prostate.The score range is 0-156 points. The higher the score is, the higher the quality of life of the subjects is. | 6 months
  The Fact-P is the Functional Assessment of Cancer Therapy-Prostate.The score range is 0-156 points. The FACT-P scale has a uniform calculation formula, which is obtained by summing up the scores of each subscale.FACT-P Total score=(PWB score)+ (SWB score) +(EWB score) + (FWB score) + (PCS score)。The higher the score is, the higher the quality of life of the subjects is.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China